CLINICAL TRIAL: NCT06368908
Title: Transcutaneous Functional Magnetic Muscle Stimulation in Critically Ill
Acronym: FMS_ICU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: General and Teaching Hospital Celje (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6I/2023/3
Record Dates: First submitted 2024-04-09; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Critical Illness Myopathy
Keywords: Critical illness; ICU acquired weakness; Functional magnetic stimulation
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: One of legs is randomised to be stimulated by trans-cutaneous functional magnetic stimulation (Arm 1), the other leg is control (Arm 2)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcutaneous functional magnetic muscle stimulation (Experimental): Transcutaneous Functional Magnetic Stimulation (FMS) Peripheral neuromuscular system stimulation will be conducted for the quadriceps femoris muscle using a magnetic stimulator (Tesla stym, Iskra Medical, Otoče, Slovenia). For magnetic stimulation, we will use pulse trains (20-50 Hz) with intensities ranging from 0.5 to 2.5 Tesla. The stimulation trains will be up to 3-6 seconds long, and the duty cycle will be varied from 1:1 to 1:10. Muscles will be stimulated with a magnetic field intensity that triggers visible contraction. The stimulation will last for 55 minutes per selected limb and will be performed 5 days a week.
  Interventions: Device: Transcutaneous Functional Magnetic Muscle Stimulation
- Control (No Intervention): the quadriceps femoris muscle of the control leg will not be stimulated by Transcutaneous Functional Magnetic Stimulation

INTERVENTIONS:
Device: Transcutaneous Functional Magnetic Muscle Stimulation — Peripheral neuromuscular system stimulation will be conducted for the quadriceps femoris muscle using a magnetic stimulator (Tesla stym, Iskra Medical, Otoče, SLO). For magnetic stimulation, we will use pulse trains (20-50 Hz) with intensities ranging from 0.5 to 2.5 Tesla. The stimulation trains will be up to 3-6 seconds long, and the duty cycle will be varied from 1:1 to 1:10. Muscles will be stimulated with a magnetic field intensity that triggers visible contraction. The stimulation will last for 55 minutes per selected limb and will be performed 5 days a week.
  Arms: Transcutaneous functional magnetic muscle stimulation

SUMMARY:
ICU-Acquired weakness (ICU-AW) is a significant complication of critical illness. ICU-AW is common in patients with sepsis, systemic inflammatory response, and mechanically ventilated. It is estimated that around 50% of patients recovering from the primary illness remain in intensive care with characteristic muscle weakness. This leads to dependence on mechanical ventilation, prolonging costly intensive care hospitalization. The myopathy causes persistent functional impairment, endangering patients long after hospital discharge.

Magnetic stimulation prevents inactivation atrophy of skeletal muscles, as demonstrated in the mobilized limb of rats. Transcutaneous magnetic stimulation of the quadriceps via the femoral nerve is a safe and painless method even when applied to humans.

In patients with chronic obstructive pulmonary disease (COPD), quadriceps magnetic stimulation increased spontaneous contraction force compared to the control group and improved quality of life. Patients with COPD tolerate quadriceps magnetic stimulation well, as it does not affect oxidative stress in muscles but does increase the size of slow-twitch muscle fibers.

In intensive care medicine, magnetic stimulation has been primarily used for diagnostic purposes in assessing diaphragm function, peripheral muscle strength assessment, and transcranial electrical stimulation as a diagnostic tool and therapeutic stimulation of brain cells. With the development of modern transcutaneous magnetic stimulators, the possibility arises for their use in intensive care medicine for therapeutic purposes such as preventing critical illness myopathy.

To date, no research has been conducted on the use and effectiveness of magnetic stimulation of peripheral muscles in critically ill individuals.

The aim of the study is to investigate the effect of Functional Muscle Magnetic Stimulation (FMS) on the development of ICU-AW.

DETAILED DESCRIPTION:
1. Introduction

   ICU-Acquired weakness (ICU-AW) is a significant complication of critical illness. ICU-AW is common in patients with sepsis, systemic inflammatory response, and mechanically ventilated. It is estimated that around 50% of patients recovering from the primary illness remain in intensive care with characteristic muscle weakness. This leads to dependence on mechanical ventilation, prolonging costly intensive care hospitalization. The resulting myopathy causes persistent functional impairment, endangering patients long after hospital discharge.

   1.1 Pathophysiological basis of development of Critical illness myopathy The pathophysiological mechanisms of ICU-AW are poorly understood, leading to the absence of specifically targeted treatments for its prevention. In most patients, skeletal muscle atrophy is observed, particularly the loss of fast-twitch muscle fibers (type II) and decreased levels of myosin heavy chains (MyHC). The loss of MyHC is a consequence of disrupted balance between its synthesis and degradation. The most significant contributors to the development of ICU-AW include systemic inflammation, sepsis, immobilization, sedation, hyperglycemia, exposure to neuromuscular blocking agents and corticosteroids, resulting in decreased muscle mass and strength. The principal intracellular system for protein degradation in skeletal muscles is the ubiquitin-proteasome system, which also regulates MyHC degradation.

   1.2 Physiotherapy and Transcutaneous Electrical Muscle Stimulation Therapeutic activity in the intensive care unit often begins with passive mobilization, especially in inactive and unconscious patients. In the treatment of critically ill patients is aimed to reduce sedation, providing appropriate analgesia, thus promoting faster awakening and cooperation, and encouraging active movement even in patients on mechanical ventilation.

   For muscle strengthening and reducing atrophy, physiotherapy is often combined with peripheral transcutaneous electrical stimulation of skeletal muscles. With electrical stimulation muscle strength can be increase in non-critically ill patients by using stimulation protocols that do not induce muscle fatigue.

   Electrical stimulation can also alter muscle functionality by decreasing the proportion of fast, glycolytic fibers (type II), which are predominant in less active individuals with predominantly sedentary lifestyles, in favor of more endurance-oriented, slow-contracting muscle fibers (type I) (fast-to-slow-transition). These changes depend significantly on the selected stimulation parameters, stimulation duration, and muscle innervation. Similarly, in critically ill patients, two consecutive skeletal muscle biopsies performed between the 5th and 15th day of hospitalization revealed a significant decrease in endurance, slow-contracting fibers.

   Electrical stimulation is a promising method for preventing critical illness myopathy, but it has certain limitations. Studies have not demonstrated its effectiveness in critically ill patients when started within the first seven days of treatment and have not been effective in very acute conditions. Electrical stimulation can induce intense and visible muscle contractions in only 75-80% of critically ill patients, possibly due to tissue edema over the muscles acting as insulation, as the depth of electrical stimulation is limited. Furthermore, electrical stimulation is a painful method, and pain assessment is more challenging in critically ill patients compared to the general population. Therefore, the selection of parameters used in muscle electrical stimulation in critically ill patients is extremely important.

   To accurately assess the effectiveness of electrical stimulation, muscle thickness assessment using ultrasound and muscle strength assessment using manual muscle testing are employed. The most common scale used for muscle strength assessment is the Medical Research Council (MRC) scale, where less than 48 points out of a maximum of 60 points or an average score of less than 4 define ICU-AW. ICU-AW encompasses both neuro- and myopathy in critically ill patients.

   Biphasic symmetric electrical stimulation with a frequency between 30-40 Hz, pulse duration of 0.3 msec, with 6 sec on and 6-12 sec off, and a total duration of 45-55 minutes has been shown to be the most effective. Patients who received electrical stimulation in addition to standard rehabilitation treatment had significantly greater muscle strength according to the MRC scale compared to patients who did not receive electrical stimulation. Moreover, we observed significantly shorter weaning from mechanical ventilation in patients who underwent muscle electrical stimulation.

   1.3 Transcutaneous Functional Muscle Magnetic Stimulation Transcutaneous Functional Muscle Magnetic Stimulation (FMS) differs from electrical stimulation in that it utilizes a magnetic applicator instead of two (or more) electrodes for muscle tissue stimulation and is significantly less painful. An electric coil installed in the applicator generates a magnetic field that propagates into space. The magnetic field also penetrates the human body, where it induces electric currents. These induced currents are electrical stimuli that, much like electrical stimulation, artificially propagate a signal along a nerve cell (neuron) and thereby cause muscle contraction. Despite the same triggering mechanism of the electric signal in the nerve cell, the method of energy delivery differs. Thus, FMS is not limited to acting solely on surface structures, which is one of the main drawbacks of electrical stimulation, as it rarely reaches structures deeper than 12 mm [38]. Unlike electrical stimulation, FMS penetrate deep into the body without direct contact of the applicator with the skin, allowing magnetic stimulation to be performed even through clothing, bandages, or on injured or sensitive skin. Additionally, in favor of FMS, it does not cause a high concentration of electric current at the point of entry into the body through the skin, hence causing no pain.

   FMS prevents inactivation atrophy of skeletal muscles, as demonstrated in the mobilized limb of rats. Transcutaneous FMS of the quadriceps via the femoral nerve is a safe and painless method even when applied to humans. At a stimulation frequency of 30Hz and a magnetic field of 1.6 T, it is capable of generating approximately 72±5% of the maximal spontaneous contraction force of the quadriceps. In patients with COPD, quadriceps FMS increased spontaneous contraction force by 17% compared to the control group and improved quality of life. Patients with COPD tolerate quadriceps FMS well, as it does not affect oxidative stress in muscles but does increase the size of slow-twitch muscle fibers.

   In intensive care medicine, magnetic stimulation has been primarily used for diagnostic purposes in assessing diaphragm function, peripheral muscle strength assessment, and transcranial electrical stimulation as a diagnostic tool and therapeutic stimulation of brain cells. With the development of modern transcutaneous magnetic stimulators, the possibility arises for their use in intensive care medicine for therapeutic purposes such as preventing critical illness myopathy. To date, no research has been conducted on the use and effectiveness of magnetic stimulation of peripheral muscles in critically ill individuals.

   1.4 Diagnosis of ICU-AW Currently, there is no single standardized diagnostic criteria to confirm the presence of ICU-AW. Clinically, muscle strength is assessed in lightly sedated participating patients. To raise suspicion of ICU-AW, clinical assessment of muscle strength is commonly performed using a modified MRC scale. This involves manual muscle testing, assessing shoulder abduction, elbow flexion, and wrist extension for upper limbs, and hip flexion, knee extension, and ankle dorsiflexion for lower limbs. The maximum total score of all assessments is 60. A score of 48 or less, or an average score of less than 4, may raise clinical suspicion of ICU-AW and associated complications. Confirming the existence of ICU-AW often requires the use of invasive diagnostic techniques such as electromyography, electroneurography, and histomorphological and molecular biological analyses of muscle and nerve biopsy samples. These techniques are considered the gold standard for diagnosis. Muscle and nerve biopsies can reveal structural anomalies, although these procedures are quite invasive and do not always provide a definitive diagnosis for ICU-AW; nevertheless, they are crucial in identifying muscle atrophy. It was demonstrated through muscle biopsy that patients with clinical and electrophysiological patterns of ICU-AW often exhibit myopathic changes. Muscle biopsies for demonstrating ICU-AW are most commonly taken from the deltoid muscle or the lateral head of the quadriceps femoris muscle [23].
2. Purpose of the study

The purpose of the study is to investigate the effect of FMS on the development of ICU-AW. The main objectives of the proposed research are:

1. To evaluate the feasibility of FMS in critically ill patients.
2. To assess the effectiveness of FMS in preventing atrophy and weakness of skeletal muscles in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* consecutive critically ill patients, already after 2 to 3 days of treatment in the ICU, whose treatment is expected to require at least 10 days in the intensive care unit.

Exclusion Criteria:

* Patients under 18 years of age
* Patients with implanted electrical devices affected by magnetic fields
* Patients with expected survival of less than 5 days
* Pregnant women
* Patients with bone and tissue injuries in the legs where standard physiotherapy cannot be performed
* Patients receiving high-dose corticosteroids (equivalent to >300 mg hydrocortisone per day)
* Patients receiving muscle relaxants
* Patients whose relatives/caregivers do not provide written consent for participation in the study
* Patients with extreme obesity (BMI over 35 kg/m2) or cachexia (BMI less than 20 kg/m2 or loss of 5% Body weight over 12 months):
* Patients with brain death
* Patients who do not consent to participate in the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-12-08 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Measurement of Thickness of Thigh Muscles | 0 day, 3-5 days, 9-12 days
  Measurement of Thickness of Thigh Muscles by Ultrasound
  Thickness and cross-section of the muscle, muscle structure, assessment of subcutaneous edema will be evaluated using ultrasound examination with a linear probe 8-12MHz (UZ apparatus Vivid 70, GE Health care, USA). Ultrasound apparatus settings (frequency 12 Hz, Gain: 55 dB, Dynamic range: 75) will be kept constant for all patients, with depth adjusted only in the case of larger muscles. Measurements will be performed in transverse and sagittal muscle sections without and with compression of the ultrasound probe.

SECONDARY OUTCOMES:
Measurement of Thigh Circumference | 0 day, 3-5 days, 9-12 days
  On the thighs, we will mark transverse and longitudinal measurement points located at the lower 1/3 of the distance between the spino-iliac point and the midpoint of the patella. The circumference of the thigh on both legs will be measured three times (first: upon enrollment in the study; second: between days 3-5 after enrollment; and third: between days 9-12 after enrollment).
Assessment of Muscle Strength and Communication Ability | at admission and at the end of study (9-12day)
  If the patient is capable of meaningful communication (Ramsay sedation scale: 2 or 3 points), the muscle strength of the upper and lower limbs will be recorded using the recommendation and scale of the Medical Research Council of Great Britain (MRC).
  On MRC scale sum of less than 48 points out of a maximum of 60 points or an average score of less than 12 ponts in 4 defined parts of the body are criteria for ICU-AW. MRC scale value of left and right leg will be compare. Lower MRC value is related to less muscle strength.
Body composition measurement by bioimpedance- Extracellular water | 0 day, 3-5 days, 9-12 days
  Body composition of the right and left body part will be assessed by bioimpedance (Bodystat, USA). Extracellular water (%, litres) will be compared between left and right body part.
Body composition measurement by bioimpedance- Intracellular water | 0 day, 3-5 days, 9-12 days
  Body composition of the right and left body part will be assessed by bioimpedance (Bodystat, USA). Intracellular water (%, litres) will be compared between left and right body part.
Body composition measurement by bioimpedance- skeletal muscle mass | 0 day, 3-5 days, 9-12 days
  Body composition of the right and left body part will be assessed by bioimpedance (Bodystat, USA). Skeletal muscle mass (kg) will be compared between left and right body part.

CONTACTS AND LOCATIONS:
Overall Officials: Roman Parežnik, MD PhD, Study Chair — General Hospital Celje
Locations (1):
- General Hospital Celje, Celje, Slovenia